CLINICAL TRIAL: NCT06004739
Title: Antibiotics for Delirium in Older Adults With No Clear Urinary Tract Infection
Acronym: A-DONUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Sault Area Hospital (Other); Michael Garron Hospital (Other); Unity Health Toronto (Other); The Ottawa Hospital (Other); Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO 4466
Record Dates: First submitted 2023-07-24; First posted 2023-08-22 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Infectious Disease
Keywords: Delirium; Antibiotics; Older adults; Urinary Tract Infection
MeSH Terms: conditions — Communicable Diseases; Delirium; Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics (Other): Participants will be randomized to start or continue with antibiotics. Antibiotic type and duration targeted to lower urinary tract infection as directed by the Most Responsible Physician (MRP).
  Interventions: Drug: Start Antibiotics / Continue Antibiotics for treatment of bacteriuria
- No Antibiotics (Other): Participants will be randomized to no antibiotics
  Interventions: Other: No Antibiotics for treatment of bacteriuria

INTERVENTIONS:
Drug: Start Antibiotics / Continue Antibiotics for treatment of bacteriuria — Participants will be randomized to start or continue with antibiotics (with antibiotic duration determined by the Most Responsible Physician [MRP]). Antibiotics choice to be selected by the MRP.
  Arms: Antibiotics
Other: No Antibiotics for treatment of bacteriuria — Participants will be randomized to no antibiotics
  Arms: No Antibiotics

SUMMARY:
Delirium is an acute confusional state that is experienced by many older adults who are admitted to hospital. To treat delirium the underlying cause needs to be identified promptly, but this is challenging. One of the potential causes of delirium is infection. Urine tests show that most patients experiencing delirium have bacteria in their urine, however, bacteria in the urine is common among older adults, and does not automatically indicate an infection is present. As a result it is difficult to know whether a lower urinary tract infection is present as individuals with delirium are frequently unable to report clinical signs of infection - symptoms of pain or discomfort with urination, having to urinate more frequently or pelvic discomfort. Very often, individuals with delirium are treated with antibiotics despite the fact that it is unknown whether antibiotics help to improve delirium in cases where bacteria in the urine is present. This proposed study is a randomized controlled trial that will examine if adults (age 60 or older) with delirium and suspected infection benefit from taking antibiotics.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 60 and admitted to a hospital ward (including rehabilitation hospital);
* Active delirium (defined by CAM: [1] inattention AND [2] acute and fluctuating level of consciousness, and either [3] disorganized thinking OR [4] altered mental status; OR physician's diagnosis)
* Less than 24 hours of antibiotics (prior to trial assessment)
* Either pyuria (defined as white blood cells detected on urinalysis or dipstick) or bacteriuria (defined as bacteria growing on urine culture)

Exclusion criteria

* Fever (temperature > 37.9C or > 100.2F) in the past 48 hours;
* Signs of lower urinary tract infection symptoms (such as new dysuria) or upper urinary symptoms (such as costovertebral tenderness)
* In the opinion of the treating physician, there is a reason apart from delirium and urine test results to treat with antibiotics (e.g., pneumonia)
* Indwelling urinary catheter for > 72 hours
* Receipt of an antibiotic where a single dose suffices for the treatment of a UTI (such as Fosfomycin)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2024-05-18 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Delirium at day 7 or at day of hospital discharge, whichever is earliest | Delirium will be assessed at the first of day 7 or discharge
  Delirium will be assessed using Confusion Assessment Method (CAM). CAM assesses 4 delirium features: [1] inattention, [2] acute and fluctuating level of consciousness, [3] disorganized thinking and [4] altered mental status. For a diagnosis of delirium by CAM, the patient must display feature [1] AND [2], AND EITHER [3] or [4].

SECONDARY OUTCOMES:
Length of hospitalization | Up to 30 days
Number of participants with bacteremia (bacteria isolated in blood culture) | Up to 7 days
Number of participants who were transferred to Intensive Care Unit (ICU) | Up to 7 days
Number of participants who had a fall | Up to 7 days
Number of participants who were physically restrained | Up to 7 days
Number of participants who received antipsychotics | Up to 7 days
Days of antibiotics | Up to 7 days
Number of participants with C. difficile infection | By 30 days
  C. difficile will be defined as a combination of a positive microbiological test for C. difficile (if still hospitalized at the time of diagnosis), or self-reported diagnosis of C. difficile (provided the patient reported diarrhea and receipt of an antibiotic to treat C. difficile)
Number of participants who died | By 30 days
Number of participants who died | By 365 days
Number of participants who were readmitted to hospital | By 365 days
Number of participants who were readmitted to hospital | By 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fralick, MD, PhD, Principal Investigator — Sinai Health System; Chris Kandel, MD, PhD, Principal Investigator — Michael Garron Hospital; Nathan Stall, MD, PhD, Principal Investigator — Sinai Health System
Locations (7):
- Northwestern Memorial Hospital, Chicago, Illinois, United States
- Canada (6):
  - The Ottawa Hospital Civic Campus, Ottawa
  - The Ottawa Hospital General Campus, Ottawa
  - Hennick Bridgepoint Hospital, Toronto
  - Michael Garron Hospital, Toronto
  - Mount Sinai Hospital, Toronto
  - Toronto General Hospital, Toronto

IPD SHARING:
Plan to Share IPD: No